CLINICAL TRIAL: NCT04187859
Title: A Feasibility Cluster RCT Investigating Improving Fluid Intake in Community-dwelling Urinary Catheterised District Nurse Patients Using an Innovative Prompting Cup, Education or a Combination of These Interventions.
Brief Title: Prompting And encouRaging Community Hydration Through EDucation
Acronym: PARCHED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cwm Taf University Health Board (NHS) (Other Government)
Collaborators: PRIME Centre Wales (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 257723
Record Dates: First submitted 2019-11-27; First posted 2019-12-05 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2019-10

CONDITIONS: Frailty
Keywords: Hydration; Fluid Intake; Frailty; Feasibility Study
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Education Session (Other): The participant will receive an education session in their home, lasting between 15-30 minutes from a District Nurse. The District Nurses will advise the participant on how to drink more fluids, the importance of hydration and the effects of dehydration.
  Interventions: Behavioral: Education Session
- Prompting Cup (Other): Participants will receive a Droplet Cup with an electronic prompting device and a brief tutorial session from the District Nurse. The Droplet Cup will encourage the participant to stay hydrated during the day, by emitting a voice or light to encourage them to drink more.
  Interventions: Device: Prompting Cup
- Control Group (No Intervention): There will be no change to the care the participant receives from the District Nurse.
- Prompting Cup and Education (Other): Participants will receive a Droplet Cup with an electronic prompting device and an education session on the importance of hydration and the effects of dehydration.
  Interventions: Behavioral: Education Session; Device: Prompting Cup

INTERVENTIONS:
Behavioral: Education Session — Participants will receive an education session from their District Nurse, advising on how to improve their hydration.
  Arms: Education Session; Prompting Cup and Education
Device: Prompting Cup — The Droplet Cup is an electronic prompting cup that emits a sound and/or light to encourage the participant to take a drink
  Arms: Prompting Cup; Prompting Cup and Education

SUMMARY:
PARCHED (Prompting And encouRaging Community Hydration through EDucation) is studying how to improve the hydration (fluid intake) of people living at home who use catheters. The investigator would like to see if improved hydration (fluid intake) reduces the risk of frailty.

PARCHED will randomise four areas in Cwm Taf University Health Board to receive one of four different interventions. Individuals will receive an intervention based on which area they live in, each participant will take part in the study for 12 weeks.

DETAILED DESCRIPTION:
PARCHED is a cluster feasibility randomized control trial (RCT) exploring the potential of an innovative prompting cup and education as person-centred and holistic tools to empower nursing leadership to reduce frailty in a catheterised community-dwelling population. This project will investigate interventions to improve hydration as potentially economically viable solutions to reducing frailty in a vulnerable population. Interventions have been developed using behaviour change theory and techniques. 80 participants will be recruited and will receive one of three interventions or usual care for a period of 12 weeks, data will be collected at baseline, 4 weeks and 12 weeks. Questionnaires, semi-structured interviews, and routine hospital records will be collected or accessed as part of the study.

ELIGIBILITY:
Inclusion Criteria:

* PARCHED will recruit district nurse patients at medium or high risk of dehydration (using the G, U and L of the GULP tool1),
* with a urinary catheter,
* living at home in community or residential care,
* aged 18 years or above

Exclusion Criteria:

* Inability to provide informed consent,
* medical conditions or dietary restrictions that would substantially limit ability to complete study requirements (i.e. intravenous fluid intake, inability to lift cup),
* living in nursing care setting,
* end of life pathway,
* diagnosed swallowing difficulty,
* inability to communicate in English or Welsh.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Recruitment of participants | 12 Weeks
Retention of participants | 12 Weeks
Retention of District Nurses | 12 Weeks
Acceptability and practicality of intervention for participants | 12 Weeks
  Participants will be approached to complete semi structured interviews which will explore the mechanisms and outcomes of the interventions.
Data Collection | 12 weeks
  Completion of Case Report Forms

SECONDARY OUTCOMES:
Hydration risk score (G, U and L of the GULP tool) | 12 weeks
Tilburg Frailty Indicator Questionnaire | 12 weeks
Fluid and food frequency questionnaires | 12 weeks
  BEV-15
Fluid and food frequency questionnaires | 12 weeks
  SSFFQ
Hydration self-efficacy Questionnaire | 12 weeks
Quality of life Questionnaire | 12 weeks
  EQ5D
PANAS mood questionnaire | 12 weeks
Montreal cognitive assessment | 12 weeks
Semi-structured longitudinal interviews with District Nurses | 12 weeks
Long-term follow up by NHS databases | 12 months
Healthcare cost questionnaire | 12 weeks
Evaluation Questionnaire | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rhian Beynon, Study Director — Cwm Taf Morgannwg University Health Board
Locations (1):
- Cwm Taf Morgannwg University Health Board, Merthyr Tydfil, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided